CLINICAL TRIAL: NCT06847269
Title: CAR T CELL Therapy for Pediatric, Adolescent and Young Adult Patients With CD19-Positive Leukemia: An Investigation of Lymphodepleting Chemotherapy Pharmacokinetics
Brief Title: CAR T CELL Therapy for Pediatric, Adolescent and Young Adult Patients With CD19-Positive Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR19PK
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; Cyclophosphamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAR19PK Therapy (Experimental): This study contains two phases.
  Collection and Manufacturing Phase:
  Patient blood cells will be collected, and possibly frozen, via a process called apheresis. These cells will then be changed to improve their ability to recognize and kill cancer cells.
  Treatment Phase:
  Patients that meet eligibility for treatment will receive lymphodepleting chemotherapy with fludarabine and cyclophosphamide, followed by an infusion of CD19-CAR T cells that were made in the Collection and Manufacturing Phase.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mesna; Biological: CD19-CAR T cell Infusion

INTERVENTIONS:
Drug: Fludarabine — Given IV
Drug: Cyclophosphamide — Given IV
Drug: Mesna — Given IV
Biological: CD19-CAR T cell Infusion — Patients will receive the CD19-CAR T cells by vein, through either an IV or a central line.

SUMMARY:
CAR19PK is a research study evaluating the use of lymphodepleting chemotherapy and chimeric antigen receptor (CAR) T cell therapy, a type of cellular therapy, for the treatment of refractory and/or relapsed leukemia. For this type of therapy, peripheral (circulating) immune cells are collected and then modified so that they can recognize an antigen, which is a particle present on the surface of a cancer cell. The CD19-CAR T cell product will be manufactured at the St. Jude Children's Research Hospital's Good Manufacturing Practice (GMP) facility.

The main purpose of this study is to determine:

* Evaluate different doses of fludarabine prior CAR T cell infusion
* How your body processes fludarabine and cyclophosphamide,
* How long the CAR T cells last in the body,
* Whether or not treatment with this therapy is effective in treating people with refractory or relapsed leukemia, and
* The side effects of this therapy.

DETAILED DESCRIPTION:
CAR19PK is a Phase II study evaluating lymphodepleting chemotherapy (age-based fludarabine dosing and cyclophosphamide), followed by infusion of CD19-CAR T cells, in pediatric and young adult patients ≤ 21 years old with relapsed/refractory CD19-positive leukemia. Treatment will include a single course of lymphodepleting chemotherapy followed by CAR T cell infusion. Lymphodepletion will include fludarabine (dosing based on age) and cyclophosphamide. The CAR T cell infusion will include a single infusion of 3x10^6 CD19-CAR T cells/kg patient weight.

This protocol contains a two-part consent process: 1) to proceed with autologous apheresis and 2) to proceed with treatment with lymphodepleting chemotherapy and infusion of the CD19-CAR T cell product.

ELIGIBILITY:
Autologous Apheresis and Manufacturing

Inclusion Criteria:

* CD19+ leukemia** with any of the following:

  * Refractory disease (primary or in relapse)
  * 2nd or greater relapse
  * Any relapse after allogeneic hematopoietic cell transplantation
  * 1st relapse if patient requires an allogeneic HCT as part of standard of care relapse therapy, but is found to be ineligible and/or unsuitable for HCT

    * must be confirmed to be CD19+ within 3 months prior to enrollment for treatment
* Age: ≤ 21 years of age
* Karnofsky or Lansky (age-dependent) performance score ≥ 50 (Appendix A)
* Estimated life expectancy of > 12 weeks. Patients with a history of prior allogeneic hematopoietic cell transplantation [HCT] must be clinically recovered from prior HCT therapy, have no evidence of active GVHD and have not received a donor lymphocyte infusion (DLI) within the 28 days prior to apheresis
* For females of child bearing age:

  * Not lactating with intent to breastfeed
  * Not pregnant with negative serum pregnancy test within 7 days prior to enrollment

Exclusion Criteria:

* Known primary immunodeficiency
* History of HIV infection
* Severe intercurrent bacterial, viral or fungal infection
* History of hypersensitivity reactions to murine protein-containing products
* Known contraindication to receiving protocol defined lymphodepleting chemotherapy regimen

Treatment

Inclusion Criteria:

* Age: ≤ 21 years of age
* Estimated life expectancy of > 8 weeks
* Detectable disease
* Prior to planned CAR T cell infusion, patients with a history of prior allogeneic HCT must:

  * be at least 3 months from HCT
  * have no evidence of active GVHD
  * have not received a donor lymphocyte infusion (DLI) within the 28 days prior to planned infusion
* Adequate cardiac function defined as left ventricular ejection fraction > 40%, or shortening fraction ≥ 25%
* EKG without evidence of clinically significant arrhythmia
* Adequate renal function defined as creatinine clearance or radioisotope GFR ³ 50 ml/min/1.73m2 (GFR ³ 40 ml/min/1.73m2 if < 2 years of age)
* Adequate pulmonary function defined as forced vital capacity (FVC) ≥ 50% of predicted value; or pulse oximetry ≥ 92% on room air if patient is unable to perform pulmonary function testing
* Karnofsky or Lansky (age-dependent) performance score ≥ 50 (Appendix A)
* Total Bilirubin ≤ 3 times the upper limit of normal for age, except in subjects with Gilbert's syndrome
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5 times the upper limit of normal for age
* Has recovered from all NCI CTAE grade III-IV, non-hematologic acute toxicities from prior therapy
* For patients of child bearing age:

  * Not lactating with intent to breastfeed
  * Not pregnant with negative serum pregnancy test within 7 days prior to enrollment
  * If sexually active, agreement to use birth control until 6 months after T cell infusion.

Exclusion Criteria:

* Active CNS-3 disease
* Known primary immunodeficiency
* History of HIV infection
* Evidence of active, uncontrolled neurologic disease
* Severe, uncontrolled bacterial, viral or fungal infection
* History of hypersensitivity reactions to murine protein-containing products
* Known contraindication to receiving protocol defined lymphodepleting chemotherapy regimen

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Fludarabine Pharmacokinetics | Days -5, -4 and -3
  Determination of Fludarabine exposure (area under the curve [AUC], mg-hr/L) using blood samples collected on days -5, -4 and -3

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Talleur, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols